CLINICAL TRIAL: NCT06179927
Title: Enhancing Theory of Mind Skills in Children With Autism Spectrum Disorder.
Brief Title: Group Intervention on Theory of Mind in Children With Autism Spectrum Disorder.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2023-008
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; children; theory of mind
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QT robot treatment (Experimental): Twenty children from the experimental group will undergo the treatment using QT Robot and the tablet.
  Interventions: Other: QT voice
- Traditional treatment (Experimental): Twenty children belonging to the control group will be subjected to the same training but in a traditional way, that is, by presenting image stimuli in a paper format.
  Interventions: Other: Image stimuli

INTERVENTIONS:
Other: QT voice — The subjects will undergo a pre-intervention assessment phase that will consist of administering the Theory Of Mind (TOM) test found in the NEuroPSYcology second edition (NEPSY) battery, part A; the same test will be re-submitted at the end of the intervention. Having ascertained the presence of the inclusion criteria and following randomization of the sample, the Experimental Group constituted of 20 children, will be administered the research task, which involves 12 sessions, one per week lasting 45 minutes. the experimental group will view 12 social scenes made via tablet. In the scenario, the depictions will be presented in color. They, guided by QT Robot's narrator voice, will have to choose from two or three alternatives the one that represents the appropriate mental state by selecting it on the tablet. Consequently, audio visual feedback will be provided, via the robot, to return information to the subject about the accuracy of the response.
  Arms: QT robot treatment
Other: Image stimuli — The subjects will undergo a pre-intervention assessment phase that will consist of administering the Theory Of Mind (TOM) test found in the NEuroPSYcology second edition (NEPSY) battery, part A; the same test will be re-submitted at the end of the intervention. Having ascertained the presence of the inclusion criteria and following randomization of the sample, the control group constituted of 20 children, will be administered the research task, which involves 12 sessions, one per week lasting 45 minutes. the experimental group will view 12 social scenes on paper. They, guided by the narrator's voice of the operator will have to choose from two or three alternatives the one that represents the appropriate mental state by indicating it on the paper. Consequently, feedback will be provided by the operator to return information to the subject on the accuracy of the response.
  Arms: Traditional treatment

SUMMARY:
The project involves the participation of 40 children with Autism Spectrum Disorder of both sexes, aged between 6 and 10 years. The subjects will undergo a pre-intervention evaluation phase, which will consist of administering the Theory of Mind (ToM) test present in the NEuroPSYcology second edition (NEPSY) battery, part A. The same test will be administered again at the end of the intervention. Once the inclusion criteria have been met and following the randomization of the sample, divided into Experimental Group (EG n=20) and Control Group (CG n=20), the administration of the search task will proceed. The study involves 12 sessions, one per week, lasting 45 minutes. The EG will view twelve social scenes created through a tablet. In the scenario, the depictions will be presented in color. Guided by the narrating voice of QT Robot, they will have to choose between two or three alternatives the one that represents the appropriate mental state by selecting it on the tablet. Consequently, an audio-visual feedback will be provided, through the robot, to give the subject information about the accuracy of their response. In both groups, a simple instruction will be given to the child, telling them to pay attention to the story that will be narrated and then answer simple questions. In the EG, QT robot will speak, while in the CG it will be the operator. The prompts will be related to the accuracy of the response or they will rather be aimed at encouraging the child to give the correct answer.

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of autism
* QS ≥ 75 assessed by administration of the GRIFFITHS scales
* Passing the emotional recognition test of the NEPSY II battery

Exclusion Criteria:

* presence of other medical disorders

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-01-22 (Estimated)

PRIMARY OUTCOMES:
NEuroPSYcology second edition (NEPSY-II) evaluations | The tests will be scheduled pre intervention (T0), at 6 months (T1) and at the study conclusion, about 1 year (T2).The test needs about 120-180 minutes.
  NEuroPSYcology second edition (NEPSY-II) is the most internationally known battery for assessing neuropsychological development in developmental age. Each NEPSY-II test provides raw scores that must be converted into scalar scores (min 1 - max 19) or percentile scores (min <2% - max >75%) according to the conversion tables in the manual. For each sub-scale higher scores correspond to better performance. NESPY's Theory of Mind (ToM) sub test, section A is used in this protocol. Assesses the ability to decode and interpret others' intentions and life points and understand how they influence behavior. the test will be given to children pre- and post-intervention.
  The ToM test is divided into verbal: the child is read scenarios or shown figures and asked questions that require understanding of the other's point of view; nonverbal: the child is asked to choose the emotional expression appropriate to the mood of a character depicted in certain contexts.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lecce S & Bianco F. Mettiti nei miei panni, Erickson 2018
- [Background] Begeer S, Howlin P, Hoddenbach E, Clauser C, Lindauer R, Clifford P, Gevers C, Boer F, Koot HM. Effects and Moderators of a Short Theory of Mind Intervention for Children with Autism Spectrum Disorder: A Randomized Controlled Trial. Autism Res. 2015 Dec;8(6):738-48. doi: 10.1002/aur.1489. Epub 2015 Apr 6. PMID 25847054
- [Background] Helen Tager-Flusberg, Evaluating the Theory-of-Mind Hypothesis of Autism, 2007
- [Background] Uta Frith, Autism and Theory of mind in everyday life, 2018